CLINICAL TRIAL: NCT05461612
Title: Initial Experience With Spatial Resynchronization Therapy in Patients With Atrial Fibrillation
Acronym: SR-TheAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxwell Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP22-001
Record Dates: First submitted 2022-07-01; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Spatial Resynchronization
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SRT Pacing (Experimental): SRT sensing and pacing of the left atrium to detect AF and restore sinus rhythm.
  Interventions: Device: Spatial Resynchronization Therapy delivered by the MAX-SRS, external recording and stimulation device

INTERVENTIONS:
Device: Spatial Resynchronization Therapy delivered by the MAX-SRS, external recording and stimulation device — Delivery of algorithmically defined pacing stimuli over a multitude of electrodes placed on the left atrium.
  Other Names: SRT, MAX-SRS

SUMMARY:
Demonstrate initial safety and performance of Spatial Resynchronization Therapy (SRT) in patients with persistent atrial fibrillation.

DETAILED DESCRIPTION:
This is an acute study to test the ability of a custom external device (MAX-SRS) to sense atrial rhythms, determine when AF is present and deliver spatial resynchronization therapy (SRT) to terminate AF.

Patients will have commercially available diagnostic electrophysiologic catheters placed in the coronary sinus and on the heart. The catheters will be connected to the MAX-SRS. If AF is not present, standard pacing measures will be used to induce AF. Once > 1 minute of AF is recorded, the MAX-SRS will be activated to sense the rhythm and deliver SRT pacing to terminate the AF. Up to five SRT deliveries using the same or different SRT algorithms will be attempted. After the first successful termination of AF or after five SRT attempts the study is complete for each patient. Diagnostic catheters will be removed after the conclusion of the SRT pacing study.

ELIGIBILITY:
Inclusion Criteria:

* Have AF that persists (Persistent AF) for more than 7 days but less than 1 year; OR has required cardioversion for termination of AF in the past 6 months; AND is not due to a reversible cause.
* Be scheduled to undergo open-heart surgery
* Be able to adhere to follow-up requirements

Exclusion Criteria:

* Have active pericarditis or any systemic infection
* Have left atrial thrombus (including left atrial appendage)
* Have had a previous attempt to ablate atrial fibrillation
* Scheduled for left atrial exclusion or excision
* Have had previous surgical intervention in the left atrium, including left atrial appendage implant or exclusion
* Have NYHA Class IV heart failure
* Have long-standing persistent or permanent AF
* Long-standing persistent AF is defined as AF that persists for greater than 1 year
* Permanent AF is defined as AF where termination (sinus rhythm) is no longer pursued
* Have any condition that prevents placement of a catheter on the posterior wall of the left atrium
* History of Left Atrium (LA) infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Ability of test system (MAX-SRS) to record AF | 60 seconds
  Record 1 run of AF = 60 seconds, categorical variable (Yes/No)
Mean SRT pacing duration per SRT pacing attempt | min:sec/attempt
  Record duration (min:sec) of each SRT pacing attempt

SECONDARY OUTCOMES:
Mean SRT pacing duration to convert AF | Mean duration (min:sec) of SRT pacing to organize clinical rhythm or terminate AF during the intra-operative procedure.
  Record duration (min:sec) of SRT pacing and organization of clinical rhythm (conversion to arrhythmia other than AF) or AF termination.

OTHER OUTCOMES:
Complications | Assessed post-procedure through hospital discharge (~7 days)
  Complications related to acute SRT pacing protocol

CONTACTS AND LOCATIONS:
Overall Officials: George Khabeishvili, MD, Principal Investigator — Tbilisi Heart and Vascular Clinic
Locations (1):
- Tbilisi Heart and Vascular Clinic, Tbilisi, Georgia